CLINICAL TRIAL: NCT01035177
Title: In Vivo Discrimination of Hip Fracture With Quantitative Computed Tomography
Brief Title: In Vivo Hip Fracture Discrimination With Quantitative Computed Tomography (QCT)
Acronym: FEMFRACT
Status: Terminated | Type: Observational
Why Stopped: Difficulties of recruitment, lack of elligible patients
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Zakia IDIR, Department Of Clinical Research of Developpement
Other Study IDs: P040404
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2008-03

CONDITIONS: Osteoporosis; Proximal Femur Fracture
Keywords: Bone Mineral Density (BMD);; Cortical bone;; Hip fracture;; Osteoporosis;; Quantitative Computed Tomography (QCT).
MeSH Terms: conditions — Osteoporosis; Proximal Femoral Fractures; Hip Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: Women without hip fracture, matched on age to the cases
- Patient: Female patients aged 60 and older with hip fracture

SUMMARY:
Numerous geometric and bone mineral density (BMD) parameters can be derived from quantitative computed tomography (QCT) images of the proximal femur analyzed using dedicated software. The primary objective is to evaluate the contribution of QCT-image analysis to the prediction of the osteoporotic hip fracture risk, as compared to the reference standard, namely, dual energy X-ray absorptiometry (DXA).

Study hypothesis: For predicting osteoporotic hip fracture, findings from QCT images of the proximal femur analyzed using dedicated software are superior over DXA measurements of proximal femoral BMD.

DETAILED DESCRIPTION:
Background Osteoporotic hip fractures exact an immense human and economic toll and therefore constitute a major public health problem. Because their incidence increases exponentially with age in both men and women, they will impose an increasing burden in the near future as the population continues to age throughout the world. In addition to the direct costs of fractures (hospitalisation and rehabilitation), the subsequent risks of death, functional impairment, dependency, and institutionalization are increased as compared to same-age individuals without fractures. Low BMD is the main risk factor for hip fracture and is generally measured using DXA, which is the reference standard.

Objectives Our research project aims to identify QCT factors that predict osteoporotic hip fracture. To this end, we will use image analysis software specially designed for proximal femur evaluation to assess 3D QCT images of the proximal femur. Femoral BMD and geometry parameters will be studied. This method has been validated experimentally. Our working hypothesis is that it will prove superior over DXA (the reference standard) in predicting osteoporotic Phip fractures.

Originality

The QCT-image analysis method investigated in our study is original, as there are no commercially available tools for measuring proximal femur BMD on QCT images. This original method grew out of 6 years of work conducted jointly at the Medical Physics Institute of the Erlangen University and the Experimental Radiology Laboratory of the LARIBOISIERE-St-Louis Research and Training Unit. Advantages of our method include 3D evaluation of the hip (with measurement of the true volumetric density), evaluation of both BMD and bone geometry, and separate evaluations of cortical and trabecular bone. DXA produces 2D images of the hip, spine, or wrist that neither provide geometric data (except projected neck length) nor allow separate analysis of cortical and trabecular bone.

We will use a case-control design to investigate postmenopausal patients with hip fracture and female age-matched controls without hip fracture.

This research project focusing on age-related bone changes is part of a multidisciplinary effort conducted by rheumatologists, radiologists, gerontologists, and orthopaedic surgeons. It will provide new information for understanding fracture pathogenesis and optimising prevention strategies in high-risk populations.

Study design We will compare geometric and BMD parameters at the proximal femur in women with PFF and in age-matched women without PFF. This is a multicenter case-control study with direct individual benefit. A diagnostic benefit exists for both the cases and the controls, who will undergo a thorough physical evaluation including routine screening for factors suggesting secondary osteoporosis, BMD measurements, and identification of risk factors for fractures (e.g., impaired balance) to allow planning of appropriate primary prevention (controls) or secondary prevention (cases). The therapeutic benefit will lie in advice regarding diet and lifestyle, calcium and vitamin D supplementation, and bisphosphonate therapy, as indicated by bone mass measurement results.

Recruitment procedure (see eligibility below)

1. Patients with PFF

   Patients with PFF will be recruited at four centres:
   * the orthopaedic surgery department of the LARIBOISIERE Teaching Hospital (Prof L. SEDEL and Prof. R. NIZARD)
   * the gerontology department at the Sainte-Périne hospital (Dr Roger)
   * the orthopaedic surgery department of the St-ANTOINE Teaching Hospital (Prof Alain SAUTET)
   * the orthopaedic surgery department of the PANTIN Center (Dr Pascal BIZOT)
2. Controls The controls will be recruited at the same four centres, either among patients referred for the diagnosis and prevention of age-related bone loss or among patients admitted for reasons other than hip fracture.

Procedures, investigations, and sample collection

1. Clinical data Age, height, weight, personal and familial medical history, smoking status, corticosteroids, treatment
2. Laboratory tests We will assay serum vitamin D levels, which are often low in women older than 65 years. All vitamin D assays for the study will be done in the same run (laboratory headed by Prof. Launay, LARIBOISIERE Teaching Hospital).
3. Bone mineral density (DXA) BMD will be measured suing a LUNAR DPX-L machine (Madison, USA). BMD measurement by DXA is the reference standard for the diagnosis of osteoporosis or osteopenia. BMD will be measured at the lumbar spine (L1 to L4) and proximal femur.
4. Quantitative computed tomography QCT allows for separate measurements in cortical and trabecular bone. Cortical bone will be evaluated at the proximal femur, and both BMD and geometry will be measured. In addition to parameters characterizing cortical bone, we will measure cancellous bone BMD and geometry. The methodology and the study parameters will vary according to the measurement site. When designing the investigation protocols, we sought the best trade-off between minimum radiation exposure and maximum image quality .

ELIGIBILITY:
Inclusion criteria:

Selection of cases: women with hip fracture

* woman aged 60 years and more
* clinical suspicion of osteoporosis based on the following: trivial trauma (fall from the standing position), history of vertebral fracture or visualization of a vertebral fracture by CT
* availability of radiographs of the proximal femur (anteroposterior view of the pelvis mandatory; anteroposterior and lateral views of the fractured hip optional)
* signature by the patient of the informed consent document

Exclusion criteria:

* patient under 60 years
* current bisphosphonate, oestrogen, or SERM treatment started more than 3 months earlier; or past treatment with these medications stopped less than 6 months earlier
* hip arthroplasty on the other side
* fracture at the site of a bone lesion
* psychiatric disorder that might prevent the patient from giving informed consent or from remaining completely still for about 15 minutes during the investigations
* informed consent document not signed by the patient

Selection of controls:

The controls will be women without hip fracture matched on age to the cases.

Inclusion criteria:

* woman aged 60 years and more
* signature by the patient of the informed consent document

Exclusion criteria:

* age under 60 years
* male
* current bisphosphonate, oestrogen, or SERM therapy started more than 3 months earlier; or past treatment with these medications stopped less than 6 months earlier
* history of osteoporotic hip fracture.
* psychiatric disorder that might prevent the patient from giving informed consent or from remaining completely still for about 15 minutes during the investigations
* informed consent document not signed by the patient

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with a history of osteoporotic hip fracture (cases) will be recruited while hospitalized in one of the study centres for immediate care of their fracture. Women without osteoporotic fractures (controls) matched on age to the cases will be recruited while receiving outpatient or inpatient care at one of the study centres. Inclusion and exclusion criteria are detailed below
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2005-02; Primary Completion 2008-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the contribution of QCT-image analysis to the prediction of the osteoporotic PFF risk, as compared to the reference standard, namely, DXA. | 1 month

SECONDARY OUTCOMES:
To compare the value of BMD parameters and geometric parameters in predicting osteoporotic PFFs | 1 month
To compare the roles for cortical bone and trabecular bone in predicting osteoporotic PFFs | 1 month
To look for differences between cervical and trochanteric hip fractures | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Valérie BOUSSON, PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Lariboisière - APHP, Paris, France